CLINICAL TRIAL: NCT07314034
Title: Facially Driven Digital Workflow for Esthetic and Functional Full-mouth Rehabilitation
Brief Title: "Facially Driven Digital Full-Mouth Rehabilitation"
Status: Recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, Clinical Professor and principle investigator, Menoufia University
Other Study IDs: ADMNF-0051
Record Dates: First submitted 2025-12-02; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Facially Driven, Fully Digital Full-Mouth Rehabilitation with Guided Implant Placement, TAD-Assisted Molar Intrusion, and Restorative Crowns/Veneers — Participants will receive full-mouth dental rehabilitation using advanced digital planning. Scans of the teeth, face, and jaw will guide treatment, which may include tooth movement with temporary devices, guided implant placement, and placement of custom veneers and crowns. This approach aims to restore bite function, improve smile esthetics, and ensure accurate, comfortable, and durable results.

SUMMARY:
Participants with bite difficulties, smile dissatisfaction, and missing mandibular molars was rehabilitated using a fully digital, facially driven workflow. Integration of intraoral, facial, and CBCT data guided esthetic design, occlusion, and implant planning, resulting in precise alignment, functional occlusion, and esthetic restoration with veneers, zirconia crowns, TAD-assisted molar intrusion, and guided implants.

DETAILED DESCRIPTION:
This Prospective study describes the comprehensive digital management of patients presenting with anterior open bite, smile dissatisfaction, and missing mandibular molars. A 3D virtual patient model was created by integrating intraoral scans, facial scans, and CBCT imaging, enabling prosthetically driven planning for esthetic and functional outcomes. Treatment involved conservative anterior rehabilitation with lithium disilicate veneers, full-coverage monolithic zirconia crowns, TAD-assisted intrusion of extruded molars, and guided implant placement for missing mandibular molars. The fully digital, facially guided workflow allowed precise restoration positioning, occlusal harmony, and predictable functional and esthetic results, demonstrating the utility of integrated digital planning in complex full-mouth rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-45 years with partial or complete edentulism requiring full-mouth rehabilitation.
* Patients with bite dysfunction, malocclusion, or esthetic concerns suitable for digital workflow treatment.
* Adequate bone volume for implant placement or candidates for TAD-assisted tooth movement.
* Willingness to undergo treatment using a fully digital, facially guided workflow and comply with follow-up visits.
* Ability to provide informed consent.

Exclusion Criteria:

* Systemic conditions contraindicating implant or surgical procedures (e.g., uncontrolled diabetes, immunosuppression).
* Active oral infections or untreated periodontal disease.
* Heavy smokers (>10 cigarettes/day) or substance abuse.
* History of head and neck radiation therapy or bisphosphonate use.
* Pregnancy or breastfeeding.
* Inability to comply with treatment or follow-up protocol.

Ages: 20 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Adult patients aged 20-45 years with partial or complete edentulism, bite dysfunction, or esthetic concerns requiring full-mouth rehabilitation. Participants must be medically fit for implant and minor orthodontic procedures, have adequate bone for implant placement or be candidates for TAD-assisted tooth movement, and be willing to undergo treatment using a fully digital, facially guided workflow. Both male and female patients capable of providing informed consent and complying with follow-up visits are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Implant Stability | 12 months post-treatment
  Clinical assessment: Absence of implant mobility assessed manually and using opposing instrument pressure.
  Radiographic assessment: Periapical radiographs using the paralleling technique to evaluate peri-implant bone levels.
  Success criteria: No progressive peri-implant radiolucency and marginal bone loss ≤ 1.5 mm during the first year, in accordance with Albrektsson et al. success criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No
Up on reasonable request